CLINICAL TRIAL: NCT01522131
Title: Treatment of Class II Furcation Defects in the Maxillary and Mandibular Molars With Bioresorbable Collagen Membrane and Laser
Brief Title: Effect of Laser Use on Guided Tissue Regeneration in Treatment of Molar Teeth With Class 2 Furcation Affected by Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Rosemary Thomas, Resident,Department of Periodontics ,School of Dentistry, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-11-0611
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-03

CONDITIONS: Furcation Defects; Periodontitis; Alveolar Bone Loss Beyond Furcation
Keywords: bioresorbable membrane
MeSH Terms: conditions — Furcation Defects; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bioresorbable membrane will be used as the control (Other): Bioresorbable membrane alone (control)
  Interventions: Procedure: bioresorbable membrane alonewill be used for regeneration of the periodontium(control)
- laser with bioresorabable membrane (test) (Experimental)
  Interventions: Procedure: bioresorbable membrane alonewill be used for regeneration of the periodontium(control)

INTERVENTIONS:
Procedure: bioresorbable membrane alonewill be used for regeneration of the periodontium(control) — bioresorbable membrane with laser will be used for regeneration of the periodontium(test)

SUMMARY:
Purpose: The proposed study will evaluate and compare the clinical response of using bioresorbable collagen membrane alone or defect debridement with erbium Laser irradiation in conjunction with bioresorbable collagen membrane in the treatment of Class II furcation defects in maxillary and mandibular teeth. The study will examine whether there is a superior regeneration potential when the laser energy is combined with membrane defect isolation.

Procedure: The study will use 2 groups, a control group and a test group with 16 patients in each group, with severe chronic periodontitis having clinical or radiographic evidence of Class II furcation defects in the buccal or lingual of the mandibular molars or Class II furcation defects on the buccal of maxillary molars. 16 patients will serve as the control group and open flap debridement with bioresorbable collagen membrane will be the mode of treatment. Group 2: 16 patients will serve as the test group and will undergo open flap debridement in conjunction with Er, Cr: YSGG laser irradiation and a bioresorbable collagen membrane will be used.

DETAILED DESCRIPTION:
All subjects will be patients of record in the Graduate Periodontics clinic at the UT School of Dentistry. These individuals will have already been diagnosed with chronic periodontitis and require surgical intervention to treat the disease process. All patients will have received initial periodontal therapy consisting of oral hygiene instructions and scaling and root planing. Once enrolled in the study, all subjects will receive surgical therapy involving opened flap debridement of the affected furcation defects along with membrane isolation of the defect. The test group will have debridement performed with the Er,Cr:YSGG laser and ultrasonic cleansing, while the control group will have hand instrumentation along with ultrasonic cleansing. This procedure will take approximately 1.5 hours. Postoperative appointments at 1,2,4,8 weeks requiring 15-30 minutes per appointment; at 3 months for periodontal maintenance and reinforcement of home care requiring 45 minutes; and at 6 months for periodontal maintenance, reassessment of the furcation defect and correction of residual defects requiring 75 minutes. Patients will be exited from the study 2 weeks after the last maintenance appointment and placed on recall with the Department of Periodontics dental hygienist. The total time commitment for each patient is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* should be 18 years of age in good general health
* should exhibit an O'Leary plaque score of 20% or less after initial therapy
* class II furcations defects should be present in the buccal of the maxillary molars or buccal or lingual of the mandibular molars
* tooth mobility should not exceed Miller Class II

Exclusion Criteria:

* patients who will be excluded include those with known hypersensitivity or allergy to chlorhexidine,
* uncontrolled diabetics,
* patients who are immunocompromised,
* who have taken steroids within 6 months of study enrollment,
* individuals who are pregnant and heavy smokers (> 10 cigarettes/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin L Weltman, DDS,MSD, Study Director — School of Dentistry ,Department of Periodontics,The University of Texas Health Science Center, Houston; Robin L Weltman, DDS,MSD, Study Chair — School of Dentistry ,Department of Periodontics,The University of Texas Health Science Center, Houston
Locations (1):
- School of Dentistry ,Department of Periodontics,The University of Texas Health Science Center, Houston, Houston, Texas, United States

REFERENCES:
- [Background] Gaspirc B, Skaleric U. Clinical evaluation of periodontal surgical treatment with an Er:YAG laser: 5-year results. J Periodontol. 2007 Oct;78(10):1864-71. doi: 10.1902/jop.2007.070054. PMID 18062108
- [Background] Crespi R, Romanos GE, Cassinelli C, Gherlone E. Effects of Er:YAG laser and ultrasonic treatment on fibroblast attachment to root surfaces: an in vitro study. J Periodontol. 2006 Jul;77(7):1217-22. doi: 10.1902/jop.2006.050416. PMID 16805685
- [Background] Pontoriero R, Lindhe J, Nyman S, Karring T, Rosenberg E, Sanavi F. Guided tissue regeneration in degree II furcation-involved mandibular molars. A clinical study. J Clin Periodontol. 1988 Apr;15(4):247-54. doi: 10.1111/j.1600-051x.1988.tb01578.x. PMID 3164333
- [Background] Lekovic V, Kenney EB, Carranza FA Jr, Danilovic V. Treatment of class II furcation defects using porous hydroxylapatite in conjunction with a polytetrafluoroethylene membrane. J Periodontol. 1990 Sep;61(9):575-8. doi: 10.1902/jop.1990.61.9.575. PMID 2170618
- [Background] Ishikawa I, Aoki A, Takasaki AA, Mizutani K, Sasaki KM, Izumi Y. Application of lasers in periodontics: true innovation or myth? Periodontol 2000. 2009;50:90-126. doi: 10.1111/j.1600-0757.2008.00283.x. No abstract available. PMID 19388956
- [Background] Derdilopoulou FV, Nonhoff J, Neumann K, Kielbassa AM. Microbiological findings after periodontal therapy using curettes, Er:YAG laser, sonic, and ultrasonic scalers. J Clin Periodontol. 2007 Jul;34(7):588-98. doi: 10.1111/j.1600-051X.2007.01093.x. PMID 17555412
- [Background] Melcher AH. On the repair potential of periodontal tissues. J Periodontol. 1976 May;47(5):256-60. doi: 10.1902/jop.1976.47.5.256. No abstract available. PMID 775048
- [Background] Darley M. Students in Sweden. Nurs Stand (1984). 1984 Nov 22;(374):8. No abstract available. PMID 6568444

RESULTS

PARTICIPANT FLOW:
Groups:
- Bioresorbable Membrane Will be Used as the Control: Bioresorbable membrane (control)
  bioresorbable membrane with laser will be used for regeneration of the periodontium: bioresorbable membrane with laser will be used for regeneration of the periodontium(test)
- Laser With Bioresorabable Membrane (Test): bioresorbable membrane with laser will be used for regeneration of the periodontium: bioresorbable membrane with laser will be used for regeneration of the periodontium(test)
Period: Overall Study
Arm/Group | Bioresorbable Membrane Will be Used as the Control | Laser With Bioresorabable Membrane (Test)
Started | 16 | 17
Completed | 14 | 17
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bioresorbable Membrane Will be Used as the Control | Laser With Bioresorabable Membrane (Test) | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Attachment( Gain or Loss) Measured by Horizontal Clinical Attachment Loss(in mm) From Baseline to 6 Months.
Description: Patients with periodontitis lose bone and clinical attachment over a period of time. In both control and test a Nabers probe( curved probe) marked in mm was used to quantify this loss or gain of clinical attachment in a horizontal direction from the cemento-enamel junction to the the most apical extent of the bone at the furcation entrance at baseline and after 6months after the procedure. These measurements were done intrasurgery and before opening of the flaps,again both at initial visit and 6 months after the procedure was done. This measurement will be measured in mm in postive numbers and then will be compared to measurements ( in mm) at intial and baseline. If there is a loss in attachment it will be denoted by negative number. If theres a gain in attachment it will be denoted by a positive number after the comparison.
Time Frame: At Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bioresorbable Membrane Will be Used as the Control | Laser With Bioresorabable Membrane (Test)
Number analyzed (Participants) | 14 | 17
mm | -.82 (1.54) | -1.26 (1.96)

2. Secondary Outcome: Clinical Evidence of Regeneration of Class 2 Furcation Defects Based on Changes in Vertical Pocket Depth Measurement(in mm)
Description: Patients with periodontitis lose bone and clinical attachment over a period of time in vertical direction also. In both control and test a UNC probe marked in mm was used to quantify this loss or gain of clinical attachment in a vertical direction from the cemento-enamel junction to the most apical extent of the bone at the furcation entrance at baseline and after 6months after the procedure. These measurements were done intrasurgery and before opening of the flaps,again both at initial visit and 6 months after the procedure was done.This measurement will be measured in mm in postive numbers and then will be compared to measurements ( in mm) at intial and baseline. Increase and decrease of vertical probing depth will be noted by a positive number.
Time Frame: At Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bioresorbable Membrane Will be Used as the Control | Laser With Bioresorabable Membrane (Test)
Number analyzed (Participants) | 14 | 17
mm | -.79 (125) | -.88 (121)

ADVERSE EVENTS:
Arm/Group | Bioresorbable Membrane Will be Used as the Control | Laser With Bioresorabable Membrane (Test)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No